CLINICAL TRIAL: NCT03019523
Title: Effects Of A Proprietary Supplement On The Acute Responses In Reaction Time, Mental Performance, And Indicators Of Focus In Athletic Populations
Brief Title: The Effect of a Caffeine Blend on Reaction Time, Mental Performance and Focus in Athletic Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mary Hardin-Baylor (Other)
Collaborators: NBTY, Inc. (Industry)
Responsible Party: Principal Investigator, Lemuel W. Taylor IV, Director, Exercise Biochemistry Laboratory, University of Mary Hardin-Baylor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NBTY-1
Record Dates: First submitted 2016-12-15; First posted 2017-01-12 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Mental Fatigue
Keywords: caffeine; mental performance; reaction time; focus
MeSH Terms: conditions — Mental Fatigue | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Maltodextrin (~2 grams to match weight of active treatment) placebo pre-testing (1 dose w/3 oz of water) 30 minutes following ingestion exercise and Makoto testing were completed.
  Interventions: Other: Sugar Pill
- Caffeine Blend (Active Comparator): 75 mg caffeine, 75 mg theanine, and 2g tyrosine pre-testing (1 dose w/3 oz of water) 30 minutes following ingestion exercise and Makoto testing were completed.
  Interventions: Dietary Supplement: Caffeine Blend

INTERVENTIONS:
Dietary Supplement: Caffeine Blend — Taken orally in capsule form
  Arms: Caffeine Blend
Other: Sugar Pill — Taken orally in capsule form
  Arms: Sugar Pill

SUMMARY:
This is a cross-over design study in which subjects arrived to the lab and were assigned a supplement to ingest. Prior to ingestion subjects completed baseline reaction time testing along with a questionnaire. Thirty minutes after ingestion subjects filled out the same questionnaire, completed a reaction time test, followed by a series of dynamic exercises. After the last exercise was finished subjects filled out the questionnaire, completed another reaction time test and repeated the series of dynamic exercises. Following the exercises, subjects filled out the questionnaire and completed a fourth round of reaction time testing. In total subjects would complete 2 rounds of dynamic exercises and 4 rounds of reaction time testing with heart rate being recorded before and after the dynamic exercise rounds. Subjects were told to wash-out for 7 days and return to the lab to complete the same testing but on the alternative supplement.

DETAILED DESCRIPTION:
Subjects expressing interest in doing the study, were interviewed in the Human Performance Lab (HPL) to determine whether they appear to qualify to participate in the study. Qualifying subjects, were then invited back to the HPL for an entry/familiarization session and be verbally told all of the requirements of the study. During this session, subjects signed Informed Consent Statements and completed personal and medical history questionnaires. Subject were familiarized to the study protocol via a verbal and written explanation outlining the study design. This included describing the testing sessions to the subjects about the tests to be performed including the Makoto testing system (reaction time testing). Subjects practiced several times during this session to eliminate the learning curve of using new equipment. Subjects were also taken through 1 round of the dynamic exercises to ensure ability to complete each exercise as needed. Subjects were then given an appointment time to perform qualifying Makoto testing to achieve greater than or equal to 70% accuracy on 3 towers at a level 7 for three consecutive trails.

Following the practice session, subjects recorded all food intake via MyFitnessPal for three days (3-d) prior to baseline testing. Subjects were instructed to refrain from exercise, caffeine, and alcohol the day prior to baseline testing and to consume their normal breakfast the morning of testing. Subjects were given a meal replacement bar in place of lunch, to consume ~2 hours before their testing session. During this time, subjects had body composition and hemodynamic assessments recorded. Two hours after ingestion of meal bar subjects reported back to the HPL and completed a Visual Analog Scale (VAS) questionnaire, a baseline Makoto prior to ingesting their assigned supplement. Thirty minutes after ingestion, Makoto and dynamic exercisers were completed. This involved subjects doing a standardized full body workout in 2 different rounds of exercise. After each round of exercise subjects filled out the VAS and performed Makoto testing. Subject then were instructed to wash-out and were scheduled for their 2nd testing session ~7 days later.

ELIGIBILITY:
Inclusion Criteria

* Subjects will be males between the ages of 18-25 years
* Subjects will be team sport athletes or highly trained
* Subjects will not be able to smoke or use tobacco
* Subjects has provided written and dated informed consent to participate in the study
* Subjects is willing and able to comply with the protocol
* Subjects is apparently healthy and free from disease, as determined by a health history questionnaire
* Subjects is a regular caffeine consumer (up to 2 cups of coffee a day)
* Subjects agrees to abstain from caffeine the day of each testing session
* Subjects agrees to abstain from exercise 24 hours prior to each testing visit. 48 hours prior to the testing session, the subject should not do anything new or unaccustomed in the form of exercise and should not increase the intensity of their workouts.

Subject Exclusion Criteria

* Subject has not been participating in regular physical activity and exercise trained for at least 12 months prior to enrollment
* Subject is diagnosed with any metabolic or chronic disease, or is on prescription medication for the diagnosed metabolic or chronic disease
* Subject is using, or has used a dietary supplement (other than a multi-vitamin/-mineral, protein powder, or meal replacements) within 6 weeks prior to enrollment. Protein/Meal Replacement Products (MRPs) must not contain any supplements such as creatine, beta-alanine, hydroxyl methlybutyrate (HMB), etc.
* Subject is in, or has participated in another clinical trial within 8 weeks prior to enrollment
* Subject has a known allergy or sensitivity to caffeine or other stimulants (determined from health history questionnaire.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Response to Caffeine on Measures of Reaction Time by Makoto | up to 4 hours
  The primary purpose of this investigation is to determine if acute ingestion of a proprietary supplement containing caffeine, theanine, and tyrosine has any positive effects on markers of reaction time in athletic populations.
Response to Caffeine on Measures of Mental Performance by Survey in Athletic Populatons | up to 4 hours
  The primary purpose of this investigation is to determine if acute ingestion of a proprietary supplement containing caffeine, theanine, and tyrosine has any positive effects on markers of mental performance in athletic populations.
Response to Caffeine on Measures of Cognitive Fatigue by Survey in Athletic Populatons | up to 4 hours
  The primary purpose of this investigation is to determine if acute ingestion of a proprietary supplement containing caffeine, theanine, and tyrosine has any positive effects on markers of cognitive fatigue in athletic populations.

SECONDARY OUTCOMES:
Response to Caffeine on Measures of Physical Performance by Comparing the Total Amount of Work Completed | up to 4 hours
  The secondary purpose of this investigation is to determine if acute ingestion of a proprietary supplement containing caffeine, theanine, and tyrosine has any positive effects on markers of physical performance in athletic populations.

CONTACTS AND LOCATIONS:
Overall Officials: Lemuel W Taylor, PhD, Principal Investigator — UMHB Human Performance Lab
Locations (1):
- UMHB Human Performance Lab, Belton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaragoza J, Tinsley G, Urbina S, Villa K, Santos E, Juaneza A, Tinnin M, Davidson C, Mitmesser S, Zhang Z, Taylor L. Effects of acute caffeine, theanine and tyrosine supplementation on mental and physical performance in athletes. J Int Soc Sports Nutr. 2019 Nov 26;16(1):56. doi: 10.1186/s12970-019-0326-3. PMID 31771598